CLINICAL TRIAL: NCT03290482
Title: Natural History of Eosinophilic Esophagitis: A Longitudinal Follow-up Over 10 Years
Brief Title: Natural History of Eosinophilic Esophagitis
Acronym: EoE
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeffrey A Alexander, Principal Investigator, Mayo Clinic
Other Study IDs: 17-002067
Record Dates: First submitted 2017-08-24; First posted 2017-09-25 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- EE Study Patients 2000-2008: All patients with the diagnosis of EE from the study period 2000 to 2008. Sixty patients participated in the 10 year follow up phone interview and questionnaire. These are the subjects we will contact to see if they are interested in participating in this study.
  If interested in participating, subjects will complete:
  1. Evaluation by the PI physical examination
  2. Complete the modified Mayo dysphagia Questionnaire (MDQ) and the Eosinophilic Esophagitis Activity Index (EEsAI) questionnaires
  3. Barium Esophagram with maximal and minimal esophageal diameter measurement
  4. EsophaCap cytology
  Interventions: Diagnostic Test: Barium Esophagram; Device: EsophaCap; Diagnostic Test: Physical Examination and Questionnaires

INTERVENTIONS:
Diagnostic Test: Barium Esophagram — Fast for 4 hours prior to the Esophagram (upper GI x-ray). You will drink a liquid that has barium or another contrast agent in it. The radiologist will use the X-ray machine to look at your upper GI tract while you drink the contrast liquid. The x-ray exam should take between 10-15 minutes.
Device: EsophaCap — Subjects will swallow the EsophaCap, which has a string attached, 10 minutes later it has devolved in the stomach. The PI will pull the string to remove the EsophaCap. We will send the sponge for cytology assessing the histologic results of eosinophils per high power field (phf)
  Other Names: Sponge
Diagnostic Test: Physical Examination and Questionnaires — Complete the modified Mayo dysphagia Questionnaire (MDQ) and the Eosinophilic Esophagitis Activity Index (EEsAI) at time of physical exam visit with PI.

SUMMARY:
Researchers are trying to understand the course of Eosinophilic Esophagitis (EoE), its progression and effects of treatments.

DETAILED DESCRIPTION:
Investigators will identify patients from their database who have been diagnosed with Eosinophilic Esophagitis (EE) from the study period 2000 to 2008, based on clinical features and biopsy findings. Participants will be offered a follow up evaluation that includes: evaluation by the Principal Investigator, completion of questionnaires, Esophagram and Esophageal sponge (EsophaCap) cytology.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older
* Previous participation in the natural history followup study

Exclusion Criteria:

* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eosinophilic Esophagitis patients that we have been following for 10 years and participated in the previous study.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Natural history of treated Eosinophilic Esophagitis (EE) | approximately 1 year
  The number of recurrent symptoms using the modified Mayo Dysphagia Questionnaire (MDQ). The MDQ is a 32 - item instrument in which symptoms are divided into three symptom domains.
Natural history of untreated Eosinophilic Esophagitis (EE) | approximately 1 year
  The number of recurrent symptoms using the modified Mayo Dysphagia Questionnaire (MDQ). The MDQ is a 32 - item instrument in which symptoms are divided into three symptom domains.
Natural history of treated Eosinophilic Esophagitis (EoE) | approximately 1 year
  The number of recurrent symptoms using the Eosinophilic Esophagitis Activity Index (EEsAI). The EEsAI provides a visual analogue of foods for subjects to examine and rate for difficulty in swallowing ranging from severe difficulties to No difficulties.
Natural history of untreated Eosinophilic Esophagitis (EoE) | approximately 1 year
  The number of recurrent symptoms using the Eosinophilic Esophagitis Activity Index (EEsAI). The EEsAI provides a visual analogue of foods for subjects to examine and rate for difficulty in swallowing ranging from severe difficulties to No difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Alexander, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cherian S, Smith NM, Forbes DA. Rapidly increasing prevalence of eosinophilic oesophagitis in Western Australia. Arch Dis Child. 2006 Dec;91(12):1000-4. doi: 10.1136/adc.2006.100974. Epub 2006 Jul 28. PMID 16877474
- [Background] Landres RT, Kuster GG, Strum WB. Eosinophilic esophagitis in a patient with vigorous achalasia. Gastroenterology. 1978 Jun;74(6):1298-1301. PMID 648822
- [Background] Fox VL, Nurko S, Furuta GT. Eosinophilic esophagitis: it's not just kid's stuff. Gastrointest Endosc. 2002 Aug;56(2):260-70. doi: 10.1016/s0016-5107(02)70188-0. No abstract available. PMID 12145607
- [Background] Straumann A, Spichtin HP, Grize L, Bucher KA, Beglinger C, Simon HU. Natural history of primary eosinophilic esophagitis: a follow-up of 30 adult patients for up to 11.5 years. Gastroenterology. 2003 Dec;125(6):1660-9. doi: 10.1053/j.gastro.2003.09.024. PMID 14724818
- [Background] Arora AS, Yamazaki K. Eosinophilic esophagitis: asthma of the esophagus? Clin Gastroenterol Hepatol. 2004 Jul;2(7):523-30. doi: 10.1016/s1542-3565(04)00236-8. PMID 15224275
- [Background] Noel RJ, Putnam PE, Rothenberg ME. Eosinophilic esophagitis. N Engl J Med. 2004 Aug 26;351(9):940-1. doi: 10.1056/NEJM200408263510924. No abstract available. PMID 15329438
- [Background] Straumann A, Simon HU. Eosinophilic esophagitis: escalating epidemiology? J Allergy Clin Immunol. 2005 Feb;115(2):418-9. doi: 10.1016/j.jaci.2004.11.006. No abstract available. PMID 15696105
- [Background] Morrow JB, Vargo JJ, Goldblum JR, Richter JE. The ringed esophagus: histological features of GERD. Am J Gastroenterol. 2001 Apr;96(4):984-9. doi: 10.1111/j.1572-0241.2001.03682.x. PMID 11316216
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials